CLINICAL TRIAL: NCT02891577
Title: Study of Ultrasonographic Cava Femoral Ratio in the Critically Ill Patient With Shock
Acronym: ECHO-RCF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: P/2015/267
Record Dates: First submitted 2016-08-11; First posted 2016-09-07 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-09

CONDITIONS: Hemodynamic Instability
Keywords: intra abdominal hypertension; shock; critically ill
MeSH Terms: conditions — Intra-Abdominal Hypertension; Shock; Critical Illness | interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Analysis of plasma creatinine, aspartate aminotransferase, and arterial blood gases.
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Ultrasonography — At the time of ICU admission, among critically ill patients with shock, the investigators will measure the diameter of the common femoral vein and that of the inferior vena cava by ultrasonography.

SUMMARY:
This study aims to describe the ratio of the diameter of inferior vena cava to the common femoral vein measured by ultrasonography in critically ill patients with shock, and to evaluate the potential link between this ratio and the existence of intra-abdominal disease.

DETAILED DESCRIPTION:
Among patients presenting with severe abdominal disease and shock, observations shown that the diameter of the common femoral vein was larger than the inferior vena cava. The hypothesis is that this observation could be secondary to a compression of the inferior vena cava related to an increased intra abdominal pressure.

ELIGIBILITY:
Inclusion Criteria:

* Adult
* Need for ICU admission
* Need for vasopressor (epinephrine or norepinephrine) to obtain a mean arterial pressure at least of 65 mmHg

Exclusion Criteria:

* Deep venous thrombosis related to inferior vena cava or common femoral veins
* Inability to measure inferior vena cava and common femoral vein diameters using ultrasonography

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients receiving catecholamine for shock state at the time of ICU admission.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-03; Primary Completion 2017-08 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Ratio of the diameter of the inferior vena cava related to the common femoral vein | Up to 28 days after ICU admission

CONTACTS AND LOCATIONS:
Overall Officials: Gaël PITON, MD, PhD, Principal Investigator — CHU Besançon
Locations (1):
- Centre Hospitalier Universitaire de Besançon, Besançon, France

IPD SHARING:
Plan to Share IPD: No